CLINICAL TRIAL: NCT06915415
Title: The Effect of Animal-Assisted Therapy on Prosocial Behavior and Emotional Regulation in Autistic Children: Comparison Between a Live Canine and a Toy Canine
Brief Title: Comparison Between a Live Canine or Toy Dog on Prosocial Behavior and Emotional Regulation in Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Michele Kilmer, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2307483365
Record Dates: First submitted 2025-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Prosocial Behavior; Emotional Regulation; Human Animal Bonding; Human Animal Interaction; Autism
Keywords: animal-assisted therapy; canine-assisted therapy; pediatric autism spectrum disorder; prosocial behavior; emotional regulation; mental health practitioners
MeSH Terms: conditions — Altruism; Emotional Regulation; Human-Animal Bond; Human-Animal Interaction; Autistic Disorder | interventions — Animal Assisted Therapy; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One group had a live canine incorporated into therapy sessions. (Experimental): The therapist included a live therapy canine to interact with participants during therapy sessions for this group. The canine is trained to provide comfort and play games with participants. Participants received cognitive behavioral therapy, sensory integration therapy, and eye movement desensitization and reprocessing therapy based upon their presenting needs. Sessions lasted between 30 to 60 minutes once weekly. Caregivers for younger participants were present throughout the session while caregivers for adolescent children were able to attend the entire session, watch the session from a different room, or stay in the lobby and meet with the therapist and participant for the last 10 minutes of therapy to review the session and therapeutic strategies to incorporate throughout the week to address deficits in emotional regulation and prosocial behavior. Sessions lasted 6 to 8 weeks, and participants could re-enroll if they desired to continue therapy to address identified concerns.
  Interventions: Behavioral: Animal-assisted therapy
- One group had a toy plush dog incorporated into therapy sessions. (Experimental): The therapist included a toy plush dog to interact with participants during therapy sessions for this group. Participants received cognitive behavioral therapy, sensory integration therapy, and eye movement desensitization and reprocessing therapy based upon their presenting needs. Sessions lasted between 30 to 60 minutes once weekly. Caregivers for younger participants were present throughout the session while caregivers for adolescent children were able to attend the entire session, watch the session from a different room, or stay in the lobby and meet with the therapist and participant for the last 10 minutes of therapy to review the session and therapeutic strategies to incorporate throughout the week to address deficits in emotional regulation and prosocial behavior. Sessions lasted 6 to 8 weeks, and participants could re-enroll in the live canine group if they desired to continue therapy to address identified concerns.
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Animal-assisted therapy — One group had a live therapy canine included in therapy sessions who was trained to provide comfort measures and promote interaction with autistic children. He is a certified therapy and service dog and knows over 50 commands and is certified in 10 autism service dog tasks. Participants played with him at the beginning of the session. They could choose to play fetch or hide and seek. Participants could say commands to make him do tricks and give him a treat as a reward. The canine would lay at participants' feet while the therapist was working on a skill in the clinic room. The canine would alert to the onset of anxiety and provide comfort measures. Participants could also cue the canine to provide comfort measures or could brush his fur and give him water as a prosocial behavior. Participants ended sessions with either fetch, soccer, or hide and seek.
  Arms: One group had a live canine incorporated into therapy sessions.
Behavioral: Behavioral therapy — One group had a toy plush dog included in therapy sessions. The therapist would incorporate the toy plush dog in the seated portion of the session to practice social skills. Participants could brush the toy plush dog, pet it, and hold it during sessions.
  Arms: One group had a toy plush dog incorporated into therapy sessions.

SUMMARY:
This study investigated the human-animal interaction (HAI) and bond (HAB) between a canine trained in therapy techniques or a canine plush toy and youth with autism spectrum disorder (ASD) during animal-assisted therapy (AAT) sessions. The purpose of this study is to explore identified gaps in knowledge pertaining to AAT in pediatric ASD care management by documenting human interaction between either a live canine or the plush toy canine during AAT sessions and evaluating prosocial behaviors observed during and after AAT sessions.

This study addressed the following research questions:

1. How do children with autism ages 2 to 18 years interact with a live canine during AAT sessions?
2. How do children with autism ages 2 to 18 years interact with a toy plush dog during AAT sessions?
3. Is there a difference in HAI in the live canine group and the toy plush dog group?
4. Is there a difference in prosocial behavior observed during AAT sessions between the live canine group and the toy plush dog group?
5. Is there a difference in behavior after AAT sessions between the live canine group and the toy plush dog group? Participants were randomly assigned to either the live canine or toy plush dog group. Adaptive functioning and social responsiveness evaluations were obtained to compare baseline behavior between the two groups. Participants attended an AAT session once weekly for 6 to 8 weeks. Each group received the same therapy provided by the therapist; the only difference being the incorporation of a live canine during the therapy session. Caregivers completed a weekly assessment depicting participants' positive and negative affect at the beginning of each session. Caregivers also completed a monthly assessment noting strengths and difficulties in social functioning and behavior at the start of the first, middle, and final session. AAT sessions were recorded and behavior occurring during the sessions was coded to note HAI and HAB that occurred during the sessions.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of autism spectrum disorder, developmental delay, or behavioral concerns.

Exclusion Criteria:

* Fearful of canines
* Allergic to canines

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of targets of interaction initiated by participants during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Targets of interaction is defined by the object or person with whom the primary participant directly interacts during AAT sessions. Participants can vocalize or verbalize, touch, make nonverbal communication, look, show affection, or demonstrate prosocial behaviors toward the target. Targets include caregivers, the therapist, the trained canine, and plush toy canine. Caregivers are defined as the participant's legal guardian or representative over age 16 years who was present during AAT sessions. Caregivers include foster parents, adoptive parents, biological parents, or extended family members such as grandparents, aunts, or uncles with whom the participant resides. The therapist is the canine handler and therapist who is conducting the sessions. The canine is a certified therapy and service dog trained to interact with autistic children. The control object is a large plush toy canine that looked and was dressed as the therapy canine and was a control condition in the study.
Number of human interactive behaviors initiated by participants during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Every instance of Social Communication or interactive behavior must engage a target (person, canine, or object). Interactive behaviors that occur between the primary participant and another person (caregiver or therapist) are considered Social Communication. Social Communication can be spontaneous or triggered by the initiation of another person. Interactive behaviors that occur between the primary participant and the canine or control object are considered Environmental Interactions. Subdomains include Talk, Gestures, Look, Touch, Affection, and Prosocial.
Number of social communication interactions initiated by participants during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interactive behaviors that occur between the primary participant and another person (caregiver or therapist) were considered Social Communication. Social Communication could be spontaneous or triggered by the initiation of another person. Subdomains include Talk, Gestures, Look, Touch, Affection, and Prosocial.
Number of environmental interactions initiated by participants during AAT sessions | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interactive behaviors that occur between the primary participant and the canine or control object are considered Environmental Interactions. Subdomains in Talk, Gestures, Look, Touch, Affection, and Prosocial.
Emotional Displays | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Emotional displays can be captured by assessing the facial expression and/or verbal content of the primary participant. Emotional display codes include Facial Emotional Display such as Smiling and Laughing, Negative Displays, No Display, or Obscured, indicating displays were not codable because they are obscured on the camera. Emotional display codes are not mutually exclusive, as many can occur within the same 10-second coding interval.
Verbal Emotional Displays | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Verbal Emotional Displays include positive, negative, or no display. This includes the content of the speech but not the tone of speech or the facial expression of the participant. If audible speech was coded under "Talk," but there are no distinguishable words, we did not code verbal emotional display. Any single statement can be coded as: (1) Positive, (2) Negative, (3) Positive and Negative, or (4) None.
Interfering Behaviors | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Interfering Behaviors coded with the OHAIRE encompass behaviors that may impair the individual's ability to participate in and benefit from an activity or interaction. These behaviors include Aggression, Overactivity, and Isolation.
Human canine interaction | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  The 3-AAT Observation ethogram was also used to code human canine interaction during AAT sessions. The revised ethogram appraises the frequency of six domains of human interaction (Affection, Play, Care, Communication, Comfort, Withdrawal) and 24 subdomains of human behavior that can occur in an AAT session. The ethogram assesses the Frequency, Intensity, and Duration of the interactions between the canine and participants.
Affection | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Affection is defined by positive behavior occurring between participants and the canine during scheduled play time incorporated into each session. Affection has two subdomains: Laughing and Petting. Intensity of Affection ranges from None (0) to Severe (4).
Laughing | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Laughing is defined as the participant laughing while playing with the canine. Audible laughter may be quiet or loud and with or without vocalization. The minimum requirement for vocalized laughter is one laugh. The minimum requirement for non-vocalized or silent laughter is two laughs with body movement such as shoulders moving to distinguish laughter from heavy breathing or sniffling.
  None (0) indicates the participant did not laugh.
  Very Mild (1) indicates the participant smiles widely showing teeth but does not audibly laugh.
  Mild (2) indicates the participant audibly once or inaudibly by moving shoulders up and down at least one time.
  Moderate (3) indicates the participant audibly two times or more or moves shoulders up and down more than twice.
  Severe (4) indicates the participant laughs more than 5 times or moves shoulders up and down more than 5 times.
Petting | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Petting is defined as the participant physically pets the canine while playing in a positive context and manner. Intensity of Petting ranges from None (0) to Severe (4).
  None (0) indicates the participant did not pet the canine during play.
  Very Mild (1) indicates the canine's skin and fur are lightly grazed when petted by participant.
  Mild (2) indicates light but clearly flush with the skin/fur of the canine. Skin and fur are lightly stretched/ shifted.
  Moderate (3) indicates more vigorous petting, fast back and forth, and skin/fur are visibly stretched/ shifted.
  Severe (4) indicates petting is very rapid, quicker back and forth, skin is very stretched, and fur is very shifted
Play | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Play is defined by the participant and canine interacting in a specific activity to promote socialization. Play has three subdomains: Fetch, Hide and Seek, and Puzzles. Intensity of Play ranges from None (0) to Severe (4).
Fetch | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Fetch is defined as the participant throwing an object, such as a ball or frisbee, in order for the canine to retrieve the object and bring the object back to the participant. This activity occurs during the scheduled play time of each session and can occur inside the clinic or outside in a grassy area in the back of the clinic. Intensity of Fetch ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play fetch with the canine.
  Very Mild (1) indicates the participant played fetch for less than 10 seconds.
  Mild (2) indicates the participant played fetch for 10-30 seconds.
  Moderate (3) indicates the participant played fetch for 30-60 seconds
  Severe (4) indicates the participant played fetch for over 60 seconds
Hide and Seek | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hide and Seek is defined as the participant playing hide and seek with the canine, either hiding themselves for the canine to find or hiding an object, such as a ball or treat, for the canine to find. This activity occurs during the scheduled play time of each session and can occur inside the clinic or outside in a grassy area in the front or back of the clinic. Intensity of Hide and Seek ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play hide and seek with the canine.
  Very Mild (1) indicates the participant played hide and seek for less than 30 seconds.
  Mild (2) indicates the participant played hide and seek for 30-60 seconds.
  Moderate (3) indicates the participant played hide and seek for 60-90 seconds.
  Severe (4) indicates the participant played hide and seek for more than 90 seconds.
Puzzles | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Puzzles is defined as the participant hiding a treat in a puzzle for the canine to solve in order to get the treat. Puzzles may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Puzzles ranges from None (0) to Severe (4).
  None (0) indicates the participant did not play puzzles with the canine.
  Very Mild (1) indicates the participant played puzzles for less than 30 seconds.
  Mild (2) indicates the participant played puzzles for 30-60 seconds.
  Moderate (3) indicates the participant played puzzles for 60-90 seconds.
  Severe (4) indicates the participant played puzzles for more than 90 seconds.
Care | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Care is defined as prosocial interactions initiated by participants to assist the canine. Care may occur during the scheduled play time or during the scheduled seated work time during the sessions. Care has two subdomains: Brush and Walking. Intensity of Care ranges from None (0) to Severe (4).
Brush | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Brush is defined by the participant using a brush to stroke the canine's coat. Brush may occur during the scheduled play time or during the scheduled seated work time during the sessions Intensity of Brush ranges from None (0) to Severe (4).
  None (0) indicates the participant did not brush the canine's coat.
  Very Mild (1) indicates the participant brushed the canine's coat for less than 30 seconds.
  Mild (2) indicates the participant brushed the canine's coat for 30-60 seconds.
  Moderate (3) indicates the participant brushed the canine's coat for 60-90 seconds.
  Severe (4) indicates the participant brushed the canine's coat for more than 90 seconds.
Walking | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Walking is defined as the participant walking the canine while holding the canine's leash. Walking may occur during the scheduled play time or during the scheduled seated work time during the sessions. Walking can occur inside the clinic or outside in a grassy area in the front or back of the clinic. Intensity of Walking ranges from None (0) to Severe (4).
  None (0) indicates the participant did not walk the canine using a leash.
  Very Mild (1) indicates the participant walked the canine using a leash for less than 30 seconds
  Mild (2) indicates the participant walked the canine using a leash for 30-60 seconds.
  Moderate (3) indicates the participant walked the canine using a leash for 60-90 seconds.
  Severe (4) indicates the participant walked the canine using a leash for more than 90 seconds.
Communication | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Communication is defined as words spoken by the participant directly to the canine. Communication may occur during the scheduled play time or during the scheduled seated work time during the sessions. Communication has three subdomains: Name, Command, and Verbal Affirmation. Intensity of Communication ranges from None (0) to Severe (4).
Name | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Name is defined as the participant saying the canine's name. Name must be directed toward the canine and not the caregiver or therapist. Intensity of Name ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say the canine's name.
  Very Mild (1) indicates the participant said the canine's name once.
  Mild (2) indicates the participant said the canine's name 2 - 3 times.
  Moderate (3) indicates the participant said the canine's name 4 - 5 times.
  Severe (4) indicates the participant said the canine's name more than 5 times.
Command | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Command is defined as the participant stating a command in order for the canine to do a trick or obey the participant. Command may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Command ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say a command.
  Very Mild (1) indicates the participant said one command.
  Mild (2) indicates the participant said commands 2 - 3 times.
  Moderate (3) indicates the participant said commands 4 - 5 times.
  Severe (4) indicates the participant said commands more than 5 times.
Verbal Affirmation | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Verbal Affirmation is defined as the participant saying verbal affirmations directed toward the canine. Verbal Affirmation may occur during the scheduled play time or during the scheduled seated work time during the sessions. Intensity of Verbal Affirmation ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say verbal affirmations.
  Very Mild (1) indicates the participant said one verbal affirmation.
  Mild (2) indicates the participant said two verbal affirmations.
  Moderate (3) indicates the participant said verbal affirmations 3 - 5 times.
  Severe (4) indicates the participant said verbal affirmations more than 5 times.
Comfort | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Comfort is defined as prosocial behavior occurring between participants and the canine. Comfort codes behavior occurring during the scheduled seated work time of each session. Comfort has ten subdomains: Head, Face, Back, Belly, Ears, Hugs, Kiss, Treat, Floor, and Laying. Intensity of Comfort ranges from None (0) to Severe (4).
Head | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Head is defined as the participant touching the top of the canine's head during seated work time. Intensity of Head ranges from None (0) to Severe (4).
  None (0) indicates the participant did not touch the top of the canine's head while seated.
  Very Mild (1) indicates the participant touched the canine's head once while seated.
  Mild (2) indicates the participant touched the canine's head twice while seated.
  Moderate (3) indicates the participant touched the canine's head 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's head more than 5 times while seated.
Face | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Face is defined as the participant touching the canine's face during seated work time. Intensity of Face ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's face while seated.
  Very Mild (1) indicates the participant touched the canine's face once while seated.
  Mild (2) indicates the participant touched the canine's face twice while seated.
  Moderate (3) indicates the participant touched the canine's face 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's face more than 5 times while seated.
Back | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Back is defined as the participant touching the canine's back during seated work time. Intensity of Back ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's back while seated.
  Very Mild (1) indicates the participant touched the canine's back once while seated.
  Mild (2) indicates the participant touched the canine's back twice while seated.
  Moderate (3) indicates the participant touched the canine's back 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's back more than 5 times while seated.
Belly | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Belly is defined as the participant touching the canine's belly during seated work time. Intensity of Belly ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's belly while seated.
  Very Mild (1) indicates the participant touched the canine's belly once while seated.
  Mild (2) indicates the participant touched the canine's belly twice while seated.
  Moderate (3) indicates the participant touched the canine's belly 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's belly more than 5 times while seated.
Ears | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Ears is defined as the participant touching the canine's ears during seated work time. Intensity of Ears ranges from None (0) to Severe (4).
  None (0) indicates the participant did not the canine's ears while seated.
  Very Mild (1) indicates the participant touched the canine's ears once while seated.
  Mild (2) indicates the participant touched the canine's ears twice while seated.
  Moderate (3) indicates the participant touched the canine's ears 3 - 5 times while seated.
  Severe (4) indicates the participant touched the canine's ears more than 5 times while seated.
Hugs | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hug is defined as the participant physically hugs the canine during seated work time. Intensity of Hug ranges from None (0) to Severe (4).
  None (0) indicates the participant did not hug the canine while seated.
  Very Mild (1) indicates the participant hugged the canine once while seated.
  Mild (2) indicates the participant hugged the canine twice while seated.
  Moderate (3) indicates the participant hugged the canine 3 - 5 times while seated.
  Severe (4) indicates the participant hugged the canine more than 5 times while seated.
Kiss | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Kiss is defined as the participant kisses the canine on his head or body during seated work time. Intensity of Kiss ranges from None (0) to Severe (4).
  None (0) indicates the participant did not kiss the canine while seated.
  Very Mild (1) indicates the participant kissed the canine once while seated.
  Mild (2) indicates the participant kissed the canine twice while seated.
  Moderate (3) indicates the participant kissed the canine 3 - 5 times while seated.
  Severe (4) indicates the participant kissed the canine more than 5 times while seated.
Treat | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Treat is defined as the participant giving the canine a treat during seated work time. Intensity of Treat ranges from None (0) to Severe (4).
  None (0) indicates the participant did not give the canine a treat while seated.
  Very Mild (1) indicates the participant gave the canine a treat once while seated.
  Mild (2) indicates the participant gave the canine a treat twice while seated.
  Moderate (3) indicates the participant gave the canine a treat 3 - 5 times while seated.
  Severe (4) indicates the participant gave the canine a treat more than 5 times while seated.
Floor | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Floor is defined as the participant sitting on the floor by the canine during the seated work time. Intensity of Floor ranges from None (0) to Severe (4).
  None (0) indicates the participant did not sit on the floor by the canine while seated.
  Very Mild (1) indicates the participant sat on the floor by the canine once while seated.
  Mild (2) indicates the participant sat on the floor by the canine twice while seated.
  Moderate (3) indicates the participant sat on the floor by the canine 3 - 5 times while seated.
  Severe (4) indicates the participant sat on the floor by the canine more than 5 times while seated.
Laying | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Laying is defined as the participant physically laying their body on the canine during the seated work time. Intensity of Laying ranges from None (0) to Severe (4).
  None (0) indicates the participant did not lay their body on the canine while seated.
  Very Mild (1) indicates the participant laid their body on the canine once while seated.
  Mild (2) indicates the participant laid their body on the canine twice while seated.
  Moderate (3) indicates the participant laid their body on the canine 3 - 5 times while seated.
  Severe (4) indicates the participant laid their body on the canine more than 5 times while seated.
Withdrawal | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Withdrawal is defined as the participant moving away from interacting from the canine. Withdrawal may occur during the scheduled play time or during the scheduled seated work time during the sessions. Withdrawal has four subdomains: Moves Away, Hides, Crying, and saying "No!" to the canine. Intensity of Withdrawal ranges from None (0) to Severe (4).
Moves Away | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Moves Away is defined as the participant physically moving away from the canine to end the interaction. Intensity of Moves Away ranges from None (0) to Severe (4).
  None (0) indicates the participant did not move away from the canine.
  Very Mild (1) indicates the participant moved away from the canine once.
  Mild (2) indicates the participant moved away from the canine twice.
  Moderate (3) indicates the participant moved away from the canine 3 - 5 times.
  Severe (4) indicates the participant moved away from the canine more than 5 times.
Hides | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Hides is defined when the participant hides their face from the canine, turns their body from the canine, or hides behind an object, such as a table, to get away from the canine. Intensity of Hides ranges from None (0) to Severe (4).
  None (0) indicates the participant did not hide from the canine.
  Very Mild (1) indicates the participant hid from the canine once.
  Mild (2) indicates the participant hid from the canine twice.
  Moderate (3) indicates the participant hid from the canine 3 - 5 times.
  Severe (4) indicates the participant hid from the canine more than 5 times.
Crying | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Crying is defined as the participant crying, with or without tears, and this behavior must be directed toward the canine. Intensity of Crying ranges from None (0) to Severe (4).
  None (0) indicates the participant did not cry with the canine.
  Very Mild (1) indicates the participant cried with the canine once.
  Mild (2) indicates the participant cried with the canine twice.
  Moderate (3) indicates the participant cried with the canine 3 - 5 times.
  Severe (4) indicates the participant cried with the canine more than 5 times.
Saying "No!" | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Saying "No!" is defined as the participant verbally stating the word "No!" to the canine to end the interaction. Intensity of "No!" ranges from None (0) to Severe (4).
  None (0) indicates the participant did not say "No!" to the canine.
  Very Mild (1) indicates the participant said "No!" to the canine once.
  Mild (2) indicates the participant said "No!" to the canine twice.
  Moderate (3) indicates the participant said "No!" to the canine 3 - 5 times.
  Severe (4) indicates the participant said "No!" to canine more than 5 times.
Frequency | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Frequency is defined by the occurrence of one of the interactions listed on the 3-AAT Observation ethogram. Interactions were measured by a tally count of each interaction.
Duration | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Duration of the interaction was assessed by rounding either up or down to the nearest 30 second mark and coded as follows.
  29 seconds or under was coded as 0.5 30 seconds to 1 minute 29 seconds was coded as 1 1:30 to 2:29 was coded as 2 2:30 to 3:29 was coded as 3 3:30 to 4:29 was coded as 4 4:30 to 5:29 was coded as 5 5:30 to 6:29 was coded as 6, and so on.
Intensity | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Intensity of the interaction was coded from None (0) to Severe (4). The mode of the interaction codes was entered to run the analysis.
Talk | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Talk is defined as verbal communication that occurs when the primary participant engages in a verbal communicative attempt with a visible target. If the target is unknown or out of frame, we coded this behavior as "No." To qualify as verbal communication, there should be audible sound clearly coming from the primary participant. We used the "three rule." If we could not determine whether the participant was talking after three viewings, we coded this behavior as "No.". If the words being spoken were intelligible, we also coded Verbal Emotional Display.
Gestures | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Gestures are defined as a form of social communication that occurs when the participant engages in a communicative attempt toward a target using physical gestures. It includes sign language and any other bodily actions that are used to communicate. The aim of the gesture should be to communicate rather than to accomplish a physical task. For example, pointing to an item on the ground is a gesture, but picking an item up off the ground is not a gesture. Talk and Gesture can be coded at the same time. When that occurred, we selected the target for BOTH codes. Gesture does not include Touch.
Look | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Look occurs when the primary participant looks in the direction of a visible target. The participant's gaze should be assessed by the angle or direction of their eyes. Look can only be coded if half of the participant's face is visible (i.e., at least one eye). Regarding canines and control objects, Look should be coded if the participant is looking at any part of the canine or object. Regarding other participants, Look can only be coded if the participant is looking at the face (or general face region) of a caregiver or therapist. If the participant looked in the direction of multiple people, canines, or objects, we coded all targets that could apply.
Touch | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Touch was coded if the primary participant comes into physical contact with a target. Touch does not include Aggression. Touch should be coded when any part of the participant's body makes contact with any part of the target. If a participant's clothing was touching another person, we also code this as Touch. Receiving any object by hand was coded as touching another person (caregiver or therapist). Similarly, receiving a control object by hand was coded as touching another person (caregiver or therapist) and the control object. In the case of giving or receiving an object by hand, we also coded this behavior as Prosocial.
Affection | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Affection was coded if the participant demonstrates physical affection or emotional warmth (i.e., verbal affection) to other humans, objects, or canines.
Prosocial | During weekly animal-assisted therapy sessions from enrollment to the end of treatment between 6 to 52 weeks
  Prosocial is defined as non-verbal behavior (i.e., physical action) that is purposefully helpful to another person, canine, or object.
Strengths and Difficulties Questionnaire | The initial SDQ is completed by caregivers at the first session (day 1) and every 4 weeks throughout the study and at the end of the study (up to 12 weeks).
  The Strengths and Difficulties Questionnaire is a behavioral screening for 2- to 17-year-olds assessing 25 attributes divided between 5 scales with values ranging from 0 to 2: Emotional Symptoms (5 items), Conduct Problems (5 items), Hyperactivity/ Inattention (5 items), Peer Relationship Problems (5 items), Prosocial Behavior (5 items). The first four domains are added together to generate a total difficulties score with values ranging 0 to 40. There are additional questions regarding the impact of the child's behavior with values ranging from 0 to 2 for a total value ranging from 0 to 10. Externalizing and Internalizing scores, values ranging from 0 to 20, are derived from the Conduct, Hyperactivity, Emotional, and Peer Problems scales. The follow-up version contains two additional items, values ranging from 0 to 4, to evaluate the perceived effect of the intervention. Higher scores in all these domains, except for the Prosocial domain, indicate problematic behavior.
Positive and Negative Affect Scale | The Positive and Negative Affect Schedule is administered at the first session of the study (day 1), and then weekly at each session throughout the study and at the end of the study (up to 12 weeks).
  The Positive and Negative Affect Schedule is a scale that consists of different words that describe feelings and emotions. The 20-item self-report assesses positive affect and negative affect. Positive affect is associated with pleasurable engagement with the environment, whereas negative reflects a dimension of general distress summarizing a variety of negative states such as anger, guilt, or anxiety. The assessment uses a 5-point scale for caregivers to select to determine if a concept applies. The final score is derived from the sum of the ten items on both the positive and negative side. Affect states include Interested, Distressed, Excited, Upset, Strong, Guilty, Scared, Hostile, Enthusiastic, Proud, Irritable, Alert, Ashamed, Inspired, Nervous, Determined, Attentive, Jittery, Active, and Afraid. Values for each item range from 1 to 5, with a total score for each affect ranging from 10 to 50. Higher scores represent higher levels of affect for each domain.
Vineland-3 | Baseline- the Vineland-3 provides baseline data of adaptive functioning and is administered within 6 months prior to Session 1.
  The Vineland, 3rd edition, is a standardized assessment measuring adaptive behavior. The overall Adaptive Behavior Composite score, with values from 20 to 160 (higher scores indicate stronger adaptive behavior) reflects scores from in three domains: Communication, Daily Living Skills, and Socialization. These three domain scores have values ranging from 20 to 115, standard score mean of 100 and standard deviation of 15, and include percentile ranks. The Vineland-3 includes optional Motor Skills and Maladaptive Behavior domains. The minimum and maximum values for the Vineland-3 Motor Skills domain are 20 and 115, with a standard score of 100 and a standard deviation of 15. Higher scores indicate fewer motor skill delays. Maladaptive Behavior domains are scored on a scale where 15 is the mean with a standard deviation of 3 points and a score greater than or equal to 18 indicates clinical significance of problematic behavior.
Social Responsiveness Scale- 2nd edition | Baseline- the SRS-2 provides baseline data of adaptive functioning and is administered within 6 months prior to Session 1.
  The Social Responsiveness Scale 2nd edition measures social ability of children from 2 years, 5 months to 18 years old. It is used primarily in research with individuals on the autism spectrum. The assessment includes a Total Score and five domain scores: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted and Repetitive Interests. It contains 65 items using a 4-point Likert scale resulting in a raw score range of 0 to 195 for the total score and 0 to 48 for each of the five treatment subscales. Higher scores reflect an increase in the occurrence of autism symptomology. The Total Score and five domain scores provide both raw scores and T-scores.

CONTACTS AND LOCATIONS:
Overall Officials: MIchele R Kilmer, DNP, Principal Investigator — The University of Arkansas
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kilmer M, Hong M, Randolph D, Reichel A, Huetter S, Bowden M, Kilmer C. Animal-assisted therapy in pediatric autism spectrum disorder: A case report. Nurse Pract. 2024 Mar 1;49(3):31-39. doi: 10.1097/01.NPR.0000000000000151. PMID 38386471
- See also: Website for the university's autism program — https://accessforautism.uark.edu/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT06915415/Prot_SAP_ICF_000.pdf